CLINICAL TRIAL: NCT02832817
Title: Accuracy and Precision of Different Devices for the Monitoring of Pulsed Oxygen Saturation
Acronym: PULSEREA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: PULSEREA2016
Record Dates: First submitted 2016-06-20; First posted 2016-07-14 (Estimated); Last update posted 2017-05-11 (Actual); Status verified 2017-05

CONDITIONS: Arterial Pulsed Oxygen Saturation
Keywords: Oxygen therapy; Pulse oximeter; Hypoxia; Hypoxemia; Arterial blood gas
MeSH Terms: conditions — Hypoxia

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Pulse oximeter — For each monitoring of Arterial Oxygen Saturation, measures of Arterial Pulsed Oxygen Saturation will be made for each pulse oximeter.

SUMMARY:
Hypoxemia is a frequent situation in clinical practice, particularly in intensive care units or perioperative. The mortality and morbidity increase for cardiovascular reason, due to hypoxia has been reported several times. It is therefore important to detect hypoxemia very early and with accuracy. The objective is to correct the causes quickly and thus avoid or minimize complications.

In addition to the risks associated with hypoxemia, the monitoring of Arterial Oxygen Saturation also avoids the adverse effects associated with hyperoxia. Indeed oxygen leads to the formation of free radicals, which in physiological condition are regulated by antioxidant mechanisms. However, in anesthesiology, it is common to find pathological situations (acute respiratory distress syndrome, shock, prolonged inflammatory state) where these regulatory mechanisms are overwhelmed. Oxygen administration to supra-physiological concentrations leads to a formation of excessive free radicals, aggravating the existing injury (including lung).

Oxygen therapy is a fully-fledged treatment requiring monitoring of its effectiveness and tolerance. Currently, the standard method for assessing oxygenation is the arterial blood gas analysis with the Arterial Oxygen Saturation. Its cost and the need for an arterial blood sample do not allow regular monitoring. Clinical evaluation of hypoxia is completely unreliable. there is a third method : monitoring devices that measure Arterial Pulsed Oxygen Saturation, called "pulse oximeters." Pulse oximeters have become an integral and mandatory part of the standard monitoring. It is through the measurement of Arterial Pulsed Oxygen Saturation, supposed to reflect Arterial Oxygen Saturation, that clinicians guide their therapeutic attitudes to optimize oxygenation and improve the prognosis of patients. So pulse oximetry is a method considered reliable and especially non-invasive. It is less expensive and does not require blood sampling. These qualities explain why these devices are easily used in anesthesia, intensive care and in emergency situations.

However, several studies have demonstrated the inaccuracy of Arterial Pulsed Oxygen Saturation in frequent situations resuscitation (shock, sepsis, dark skin type). Thus, it is necessary to objectify the benefits and limitations of pulse oximetry to optimize their use, especially in these situations of high risk, where a discrepancy between the values measured by the pulse oximetry and measurement of arterial blood saturation with oxygen gas can be detrimental.

It exists several pulse oximetry devices, whose accuracy seems unequal, which necessitates a comparative study.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in intensive care
* Over 18 years
* Continuous monitoring of oxygen saturation
* Susceptible oo have arterial blood gases and carrying an arterial catheter

Exclusion Criteria:

* patient protected by the law
* no social security number
* carbon monoxide Intoxication
* High methemoglobinemia.
* Therapeutic limitation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General population of Intensive Care Unit
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2016-02-20 (Actual); Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Oxygen saturation by pulse oximetry monitoring accuracy | at each arterial blood gas during ICU hospitalization (max 5 punctures from inclusion to ICU discharge - average of 1 week)
  determine the accuracy of oxygen saturation by pulse oximetry monitoring devices (SpO2) compared to the reference method, arterial oxygen saturation (SaO2) by blood gas on Co-Oximeter

SECONDARY OUTCOMES:
Number of participants for whom there will be mismatch between SpO2 (oxygen saturation by pulse oximetry) and SaO2 (arterial oxygen saturation) measures with medical adverse events (vasopressors, hypoxemia, acidosis, alkalosis) | at each arterial blood gas during ICU hospitalization (max 5 punctures from inclusion to ICU discharge - average of 1 week)
  highlight groups with risks of discrepancy between SpO2 and Sa02, and describe with the following criteria : presence of vasopressors, mechanical ventilation, blood lactate value, hypoxemia, acidosis / alkalosis, skin hypoperfusion signs, skin phototype, temperature.

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Réanimation Chirurgicale, Angers, France